CLINICAL TRIAL: NCT02803216
Title: Traditional Chinese Medicine Combined With Standard Triple Region for Eradication of Helicobacter Pylori: a Prospective, Double-blinded, Randomized Trial
Brief Title: Traditional Chinese Medicine Combined With Standard Triple Region for Eradication of Helicobacter Pylori
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Digestion-02
Record Dates: First submitted 2016-05-31; First posted 2016-06-16 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-06

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Omeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard triple region (Experimental): The patients in this group were given 10-day standard triple therapy.
  Interventions: Drug: standard triple region
- standard triple region +2-week TCM (Active Comparator): The patients in this group were given 10 days of standard triple therapy + 2-week Xiang-sha-liu-jun decoction.
  Interventions: Drug: standard triple region; Drug: 2-week Xiang-sha-liu-jun decoction
- standard triple region +4-week TCM (Active Comparator): The patients in this group were given 10days of standard triple therapy + 4-week Xiang-sha-liu-jun decoction.
  Interventions: Drug: standard triple region; Drug: 4-week Xiang-sha-liu-jun decoction

INTERVENTIONS:
Drug: standard triple region — ten days of standard triple region (20mg omeprazole 20mg, 1.0 amoxicillin, 0.5 clarithromycin, Bid).
  Other Names: omeprazole, amoxicillin, clarithromycin
Drug: 2-week Xiang-sha-liu-jun decoction — 2-week Xiang-sha-liu-jun decoction, bid.
  Arms: standard triple region +2-week TCM
Drug: 4-week Xiang-sha-liu-jun decoction — 4-week Xiang-sha-liu-jun decoction, bid.
  Arms: standard triple region +4-week TCM

SUMMARY:
To evaluate the efficacy and safety of Traditional Chinese Medicine (TCM) decoction and powder combined with standard triple therapy on improving eradication rate of Helicobacter Pylori (H. pylori).A multi-center randomized control clinical trial design was adopted in the trial.

ELIGIBILITY:
Inclusion Criteria:

* those who met chronic gastritis (chronic superficial gastritis and chronic atrophic gastritis) diagnostic criteria;
* aged between 18-65 years old;
* positive H. pylori infection confirmed by two or more methods of different
* principles (stop using PPI, H2RA, bismuth, and antibiotics since two weeks before examination);
* patients were informed consent and willing to accept corresponding treatments.

Exclusion criteria:

* Patients having chronic atrophic gastritis with severe dysplasia, upper gastrointestinal bleeding, peptic ulcers, and gastrointestinal tumors;
* digestive organic disease (such as chronic pancreatitis, cirrhosis, etc.), or systemic diseases affecting intestinal motility (such as hyperthyroidism, diabetes mellitus, chronic renal insufficiency, mental, and neurological diseases, etc.);
* those who were accompanied by serious heart, liver and other major organs lesions, blood diseases, and cancer (ALT, AST two times higher than normal value);
* those who had taken medicines that might affect H. pylori detection results within two weeks (antacids, H2RA, PPIs, bismuth and antibiotics, etc.);
* pregnant and lactating women; patients with history of systematic and neuropsychiatric disorders; those who had history of any drug allergy; and those who were participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | 13C or 14C urea breath test was performed at four weeks after western medicine termination.

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | at baseline, and every week up to four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: xudong Tang, Ph.D, Study Chair — XiYuan Hospital of China Academy of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Yes